CLINICAL TRIAL: NCT02082431
Title: Long QT & Hearing Loss Prospective Study Registry
Brief Title: Determine the Incidence of Long QT Amongst a Large Cohort of Subjects Diagnosed With Unilateral or Bilateral Sensorineural Hearing Loss.
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-001-13
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Sensorineural Hearing Loss; Long QT Syndrome
Keywords: Sensorineural hearing loss; Long QT Syndrome
MeSH Terms: conditions — Hearing Loss, Sensorineural; Long QT Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the true incidence of long QT (LQT) amongst a large cohort of subjects diagnosed with unilateral (right/left) or bilateral sensorineural hearing loss.

DETAILED DESCRIPTION:
The purpose of this study is to determine the true incidence of long QT (LQT) amongst a large cohort of subjects diagnosed with unilateral (right/left) or bilateral sensorineural hearing loss.

The goal of this study is to answer the following questions:

1. What is the incidence of an abnormal ECG (QTc > 450 msec) in neonates greater than a week of age with either unilateral or bilateral Sensorineural hearing loss?
2. What percentage of neonates greater than one week of age with either bilateral or unilateral sensorineural hearing loss and an abnormal ECG have an identifiable genetic mutation?
3. What is the incidence of an abnormal genetic mutation consistent with long QT regardless of the ECG in neonates with bilateral sensorineural hearing loss?

ELIGIBILITY:
Inclusion Criteria:

* All newborns who demonstrate a refer in one or both ears on a routine newborn hearing screen
* Documentation of informed consent
* Inborn
* Ability to perform an ABR (auditory brainstem response screen technology) screening test
* No major anomalies
* Subjects' parents willing to provide follow-up data on their child

Exclusion Criteria:

* Newborns with a syndromic cause of hearing loss
* Parents unwilling to provide follow-up data
* Major congenital anomalies
* Major medical problem or conditions. (i.e., hypoxic ischemic encephalopathy (HIE), persistent pulmonary hypertension neonate (PPHN), meconium aspiration, etc.)
* Congenital cytomegalovirus (CMV)

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn infants
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-08; Primary Completion 2020-02-18 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
The incidence of an abnormal ECG (QTc > 450) in neonates greater than a week of age with either unilateral or bilateral sensorineural hearing loss | 6 months
  ECG results to determine QTc length

SECONDARY OUTCOMES:
In neonates > 1 week of age with either bilateral or unilateral sensorineural hearing loss and an abnormal ECG, percentage have an identifiable genetic mutation | One year
  Audiology diagnostic results

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cohen, MD, Principal Investigator — Pediatrix
Locations (12):
- United States (12):
  - Jack Jacob, Anchorage, Alaska
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Lawrence and Memorial Hospital, Waterford, Connecticut
  - Swedish American Hospital, Rockford, Illinois
  - Hearts for Hearing, Oklahoma City, Oklahoma
  - Dell Children's Medical Center, Austin, Texas
  - Child Cardiology Associates, Austin, Texas
  - Christus Santa Rosa Westover Hills, San Antonio, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Alexandria Hospital- Inova Health System, Alexandria, Virginia
  - Pediatrix Audiology Services, Fairfax, Virginia

REFERENCES:
- [Derived] Fenrich AL, Shmorhun DP, Martin GC, Young JA, Cohen MI, Kelleher AS, Anyebuno MA, Rider ED, Motta CL, Clark RH. Long QT and Hearing Loss in High-Risk Infants Prospective Study Registry. Pediatr Cardiol. 2022 Dec;43(8):1898-1902. doi: 10.1007/s00246-022-02939-4. Epub 2022 Jun 3. PMID 35661239